CLINICAL TRIAL: NCT06697561
Title: Development and Evaluation of an Evidence-based Education Program for People With Hand Dysfunction in Scleroderma: A Randomized Control Trail
Brief Title: Development and Evaluation of an Evidence-based Education Program for People With Hand Dysfunction in Scleroderma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wen-Shao Lin (Other)
Collaborators: Cheng Hsin Rehabilitation Medical Center (Other); National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Wen-Shao Lin, Nurse Practitioner, Cheng-Hsin General Hospital
Organization: Cheng-Hsin General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: (1106)113A-36
Record Dates: First submitted 2024-11-16; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Scleroderma, Systemic
Keywords: Scleroderma; Hand dysfunction; Evidence-based knowledge translation; Patient education
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education group (Experimental): receives the "Evidence-Based Education Program for people with hand dysfunction in scleroderma" (which includes: educational handbook on self-care for hand dysfunction in scleroderma, multimedia teaching materials, and individualized consultations).
  Interventions: Behavioral: patient education program
- control group (No Intervention): Receives usual care

INTERVENTIONS:
Behavioral: patient education program — The intervention for the experimental group was an "evidence-based educational program for hand dysfunction in patients with systemic sclerosis," which included a health education manual and multimedia videos developed through evidence translation. Additionally, individual education and consultation were provided.
  Arms: Patient education group

SUMMARY:
The purpose of this study is to develop an evidence-based educational program for scleroderma patients with hand dysfunction. The program includes a self-care handbook and multimedia video resources. The study aims to answer:

Does the intervention improve hand function in the experimental group compared to the control group? Does the intervention improve self-care knowledge of hand dysfunction? Does the intervention improve overall health?

Participants will receive an 8-week program, while the control group receives usual care. Outcome measures include hand function, overall health, and self-care knowledge.

DETAILED DESCRIPTION:
The study will adopt a repeated measures randomized controlled trial design (parallel randomized controlled trial) using convenience sampling. Participants in the experimental group will receive an "evidence-based scleroderma hand dysfunction education program" provided by the researchers for eight weeks. The control group will receive standard medical care during the study period and will receive the same scleroderma hand dysfunction education program as the experimental group after the study concludes. Both groups will undergo pre-intervention assessments, as well as post-intervention assessments at the fourth and eighth weeks. The primary outcome measures include evaluating the effectiveness of the education program in improving hand dysfunction severity, overall health, adherence to rehabilitation exercises, and self-care knowledge related to hand dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with systemic sclerosis who meet the 2013 American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) diagnostic criteria and have hand dysfunction.
2. Adults aged 18 years or older.
3. Participants who are conscious and able to communicate in Mandarin Chinese or Taiwanese Hokkien.
4. Participants who provide informed consent to participate in the study after being briefed on its purpose.

Exclusion Criteria:

1. Participants who have participated in any other hand rehabilitation program within the past three months.

2, Participants with organic brain dysfunction. 3. Participants with severe visual or hearing impairments. 4. Participants with serious illnesses that hinder communication or interfere with the normal learning process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-developed questionnaire on self-care knowledge for scleroderma hand dysfunction | At baseline, 4 weeks, and 8 weeks post-intervention
  The "Scleroderma Hand Function-Related Self-Care Knowledge Scale," validated by experts for reliability and validity, consists of 15 items. The scale uses a dichotomous scoring method with three response options: "True," "False," and "Don't know." It includes both positively and negatively worded items. Correct answers are scored as one point, while incorrect answers and "Don't know" responses are scored as zero. The total score ranges from 0 to 15, with higher scores indicating a greater level of self-care knowledge regarding scleroderma-related hand function impairments.
Grip strength | At baseline, 4 weeks, and 8 weeks post-intervention.
  Grip strength of the dominant hand (in kg) will be measured using a dynamometer, and the average of three trials will be used as the final muscle strength assessment indicator.
delta finger-to-palm, Delta-FTP | At baseline, 4 weeks, and 8 weeks post-intervention.
  Delta-FTP refers to the difference in distance between the tip of the third finger and the midpoint of the distal palmar crease when the finger is fully extended and fully flexed. It is an effective measurement method to assess the range of motion and flexibility of fingers in patients with scleroderma.
Raynaud's phenomenon visual analog scale | At baseline, 4 weeks, and 8 weeks post-intervention.
  This scale evaluates the severity and impact of Raynaud's phenomenon on daily activities in patients with scleroderma over the past week. Scores range from 0 mm (no impact) to 100 mm (very severe impact), with higher scores indicating greater impairment of hand function
Digital ulcers visual analog scale | At baseline, 4 weeks, and 8 weeks post-intervention.
  This scale evaluates the severity and impact of Digital ulcers on daily activities in patients with scleroderma over the past week. Scores range from 0 mm (no impact) to 100 mm (very severe impact), with higher scores indicating greater impairment of hand function.

SECONDARY OUTCOMES:
Overall disease severity visual analog scale | At baseline, 4 weeks, and 8 weeks post-intervention
  This scale measures the patient's self-assessed overall disease severity, ranging from 0 to 100, where 0 indicates the best health and 100 indicates the worst health, with higher scores indicating poorer overall health status.
Adherence to Hand Exercise Training | At baseline, 4 weeks, and 8 weeks post-intervention.
  Using an exercise diary as an evaluation tool to assess the effectiveness of adherence to rehabilitation exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Hsin General Hospital, Principal Investigator — Institutional Review Board
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan